CLINICAL TRIAL: NCT04535492
Title: Improving Cancer Screening Through A Tailored Technology-Based Intervention
Brief Title: Technology-Based Cancer Screening Intervention
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No further funding
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Vanessa Diaz, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 00101494; 1R61AG068951 (NIH)
Record Dates: First submitted 2020-08-27; First posted 2020-09-02 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Cancer; Lung Cancer; Breast Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Lung Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Colorectal Cancer Screening Recommended (Other): The USPSTF recommends screening for colorectal cancer starting at age 50 years and continuing until age 75 years.
  Interventions: Behavioral: Decision Making Support Tool
- Lung Cancer Screening Recommended (Other): The USPSTF recommends annual screening for lung cancer with low-dose computed tomography (LDCT) in adults ages 50 to 80 years who have a 20 pack-year smoking history and currently smoke or have quit within the past 15 years.
  Interventions: Behavioral: Decision Making Support Tool
- Breast Cancer Screening Recommended (Other): The USPSTF recommends biennial screening mammography for women aged 50 to 74 years.
  Interventions: Behavioral: Decision Making Support Tool

INTERVENTIONS:
Behavioral: Decision Making Support Tool — Primary care practices randomized in a stepped wedge cluster design will implement a newly developed predictive model and analytic tool to improve shared decision-making for patients.

SUMMARY:
The primary purpose of this research study is to contribute to generalized knowledge on how to increase screening for patients at risk of missing their recommended cancer preventive care by using a newly developed predictive model and analytic tool to improve shared decision-making for these patients. The goal of the clinical trial is to evaluate (prove) the effectiveness of this shared-decision making support tool developed in EPIC on the rate of recommended cancer screening in practice. It contributes to knowledge on what specific methods can increase patient adherence to recommended preventive care and reduce disparities.

DETAILED DESCRIPTION:
Patients seen at primary care practices, who have been pre-determined to have unmet screening requirements and have received standard of care with a QI tool, will be asked to complete an optional questionnaire electronically through a patient portal or via a link sent by text within a week of their visit, based on their preference. Only those who have indicated they agree to be contacted for research purposes will be contacted. Surveys will be distributed through REDCap so no identifying information will be contained in the answers. REDCap is a free, HIPAA compliant interface for building and managing online databases. Additionally, surveys will be sent via mail if the patient cannot be reached electronically. Survey responses received through the mail will not include any identifying information. Pre-paid return envelopes will be provided to preserve anonymity. Although a small proportion of South Carolina's population are primary Spanish speakers (about 4%), to be inclusive we want to ensure all materials are available in Spanish. To remove barriers to participation, those needing physical, hearing, and visual assistance will be able to review and complete documents at the time of their clinic visit with the assistance of trained study personnel. Invitations will continue to be sent out until 100 total patient responses are received per practice in the pragmatic trial, or 50 per practice in the pilot. Clinicians will also receive a survey to assess the tool. Recruitment for clinicians surveys will be done via email sent by the practice managers to the providers who have agreed to use the QI tool. Clinician assessments will be delivered electronically via a link delivery by email or text, or sent by mail, based on clinician preference. Respondents will be reimbursed for their time and effort. These assessments will be anonymous. Survey participation will be coded in order to provide compensation. Since data will be identified only by code numbers (participant IDs) the master list of those codes will be kept physically separate from the collected data.

ELIGIBILITY:
Breast Cancer Screening:

Inclusion Criteria: women 50-74 years old Exclusion Criteria: current breast cancer diagnosis, mastectomy

Colorectal Cancer Screening:

Inclusion Criteria: adults 50-74 years Exclusion Criteria: colorectal cancer diagnosis

Lung Cancer Screening:

Inclusion Criteria: adult 55-80 years old with 30 pack per year history who currently smoke or quit within the last 15 years.

Exclusion Criteria: lung cancer diagnosis

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of successful completion of breast cancer screening noted via electronic health record having mammogram result for the patient. | Duration of the study, a total of five years.
  Successful completion rate per practice involved, based on eligible patients.
Rate of successful completion of lung cancer screening noted via electronic health record having low dose computed tomography of the chest result for the patient. | Duration of the study, a total of five years.
  Successful completion rate per practice involved, based on eligible patients.
Rate of successful completion of colorectal cancer screening noted via electronic health record having colonoscopy, fecal occult blood, or non invasive screening option result for the patient. | Duration of the study, a total of five years.
  Successful completion rate per practice involved, based on eligible patients.

SECONDARY OUTCOMES:
Average score of patient experience and satisfaction as assessed via Likert scale survey. | Duration of the study, a total five years.
  A 23 item survey with Likert scale question is used to compiled the patient response: 23 is the lowest score and represent dissatisfaction and 115 is the highest score and represent satisfaction. Participants will have the option to enter text for qualitative feedback and analysis.
Average score of clinician experience and satisfaction as assessed via Likert scale survey. | Duration of the study, a total five years.
  A 20 item survey with Likert scale question is used to compiled the patient response: 20 is the lowest score and represent dissatisfaction and 100 is the highest score and represent satisfaction. Participants will have the option to enter text for qualitative feedback and analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Diaz, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Dataverse, an open source research data repository, will be used to archive and share de-identified participant data.
Supporting Information: Study Protocol, Analytic Code
Time Frame: From the end of the study, July 2025, to July 2030.